CLINICAL TRIAL: NCT03053154
Title: Influence Of Pelvic Inclination On Sit To Stand Task In Stroke Patients
Brief Title: Relationship Between Pelvic Tilt and Sit to Stand Task in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar El-sayed Ismail, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/001363
Record Dates: First submitted 2017-01-22; First posted 2017-02-14 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Stroke
Keywords: Pelvic Inclination; Sit to Stand; Stroke; Anterior pelvic tilt; Posterior pelvic tilt
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Experimental group1: 15 stroke patients with right side affection, their age ranged form 45 to 60 were recruited to assess the pelvic tilt angles from sitting position and from the dynamic task of sit to stand.
  Interventions: Other: Sagittal pelvic tilt assessment
- Experimental group2: 15 stroke patients with left side affection, their age ranged form 45 to 60 were recruited to assess the pelvic tilt angles from sitting position and from the dynamic task of sit to stand.
  Interventions: Other: Sagittal pelvic tilt assessment
- Control group: 15 Normal subjects without any diseases or dysfunctions , their age ranged form 45 to 60 were recruited to assess the pelvic tilt angles from sitting position and from the dynamic task of sit to stand.
  Interventions: Other: Sagittal pelvic tilt assessment

INTERVENTIONS:
Other: Sagittal pelvic tilt assessment — Each group passed by three phases of assessment. Firstly assess the pelvic tilt angles from sitting position. Secondly assess the pelvic tilt angles from dynamic sit to stand task. Thirdly, assess the ability to perform sit to stand task of each participant.

SUMMARY:
The purpose of this study is to assess and determine the influence of pelvic inclination on sit to stand task in stroke patients.

DETAILED DESCRIPTION:
There is a crucial need to have a better understanding of effect of pelvic inclination on sit to stand activity and to know the important factors to be considered to improve the patients' treatment and performance. Forty five participants are recruiting to assess the pelvic tilt angles in stroke patients during sitting position and to analyze the influence of pelvic tilt angles on ability to perform sit to stand task during rising from a chair in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ranged from 45-60 years old.
* Normal body weight with a body mass index (BMI) ranged from 18.5 to 24.9 kg/m2.
* Patients' had the ability to maintain sitting position without using any aids.
* Patients' had the ability to stand from sitting five times independently.
* Cooperative patients with ability to understand instructions and follow simple verbal commands.
* The duration of illness was from six months to 2 years.
* The degree of the paretic lower limb spasticity ranged between (1:1+) according to the Modified Ashworth Scale.
* The degree of the paretic lower limb weakness was not less than grade 3 according to group muscle testing.

Exclusion Criteria:

* History of previous strokes and other neurological disorders.
* Visual, auditory and vestibular deficits.
* Cognitive impairments and language deficits.
* Leg length discrepancy is more than 0.5 cm.
* Previous history of orthopedic conditions in back or lower limbs (e.g. low back pain, fractures, deformities and surgeries).

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The patients were recruited from the Out-patient clinic for Neuromuscular Disorders and Its Surgery, Faculty of Physical Therapy, Cairo University and Out- patient clinic of El-kasr El-Aini Hospital, Faculty of Medicine, Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
posterior pelvic tilt angle | One shot (Each participant was assessed immediately and it takes about 15 minutes)
  Posterior pelvic tilt angle measured by the palpation meter (PALM) inclinometer. It was assessed as one shot in one assessment session.

SECONDARY OUTCOMES:
Pelvic Inclination analysis in sit to stand task | One shot (Each participant is assessed immediately and it takes about 10 minutes)
  Pelvic Inclination analysis in sit to stand task by Two dimensional video based motion analysis in three phases of sit to stand task. It will be assessed as one shot in one assessment session.

CONTACTS AND LOCATIONS:
Overall Officials: Manar El-sayed Ismail — Cairo University; Moshera H. Darwesh, Professor — Cairo University; Sandra M. Ahmed, Assistant Professor — Cairo University
Locations (1):
- Manar El-sayed Ismail, Giza, Egypt